CLINICAL TRIAL: NCT06287502
Title: Efficacy of Structured Exercise-Nutritional Intervention on Sarcopenia in Patients With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kowloon Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Hin Cheung, Principal Investigator, Kowloon Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHRehab_LeungHC_2
Record Dates: First submitted 2024-02-16; First posted 2024-03-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia; Osteoporosis
MeSH Terms: conditions — Sarcopenia; Osteoporosis | interventions — Pliability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Subjects received resistance, aerobic, flexibility and balance exercise training; and nutritional supplement containing β-hydroxy β-methylbutyrate (HMB) during the 12-week study period.
  Interventions: Dietary Supplement: β-hydroxy β-methylbutyrate (HMB); Behavioral: Resistance, aerobic, flexibility and balance exercise training
- Wait-list control (No Intervention): The waitlist control group would receive 12 weeks of conventional care. After the study period, they would receive the same intervention.

INTERVENTIONS:
Dietary Supplement: β-hydroxy β-methylbutyrate (HMB) — Ensure NutriVigor, a nutritional supplement, was provided to subjects according to the manufacturer's recommendation of two servings per day. Each serving consists of 54.1g of powder which provides ~231kcal, 8.61g protein, 1.21 g β-hydroxy β-methylbutyrate, 130 IU vitamin D and 0.29 g omega-3 fatty acid.
  Arms: Intervention
Behavioral: Resistance, aerobic, flexibility and balance exercise training — The exercise intervention consists of 75-minutes sessions delivered by physiotherapists at the Integrated Rehabilitation Day Centre (IRDC) in Kowloon Hospital, twice per week for 12 weeks with a total of 24 supervised sessions. Each exercise session consists of 5 minutes of warm up, 30 minutes of resistance training, 20 minutes of aerobic training, 15 minutes of balance or neuromuscular exercises and 5 minutes of cool down.
  Arms: Intervention

SUMMARY:
This is a prospective parallel group, double-blinded randomized controlled trial. Subjects are randomized into two groups - the intervention group and waitlist control group. Subjects received resistance, aerobic, flexibility and balance exercise training; and nutritional supplement containing β-hydroxy β-methylbutyrate (HMB). The intervention group would first receive the intervention during the 12-week study period. Meanwhile, the waitlist control group would receive 12 weeks of conventional care. After the study period, they would receive the same intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sarcopenia:

   * Low hand grip strength (Male: <28 kg, Female: <18 kg) AND
   * Low appendicular skeletal mass by bioimpedance analysis (Male: <7.0 kg/m2 Female: <5.7 kg/m2)
2. Diagnosed with osteoporosis by:

   * Fragility fracture or
   * T-score ≤-2.5 SDs at any site based upon BMD measurement by Dual Energy X-ray Absorptiometry (DXA) scan

Exclusion Criteria:

1. Incompetent in giving consent or following commands
2. Non-ambulatory subject
3. Unstable medical conditions contributing to sarcopenia, for example but not limited to:

   1. End stage organ failure
   2. Unstable cardiovascular, respiratory, gastrointestinal and endocrine conditions
   3. Active malignancy
4. Chronic kidney disease stage IV or above or with hyperkalaemia
5. Diabetes mellitus on medications or with unstable control
6. Terminal illness
7. Obese subjects (BMI ≥ 25.0)
8. Self-reported allergy to the ingredients of the nutrition supplement
9. Patients with metallic implants
10. Any orthopaedic pathologies affecting the strength of bilateral upper limbs
11. Any hereditary or acquired muscular diseases
12. Participation in other regular exercise programme

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Grip strength | 12 weeks
  Grip strength was measured with Jamar Plus+ digital hand dynamometer (Performance Health Supply, Wisconsin, United States).

SECONDARY OUTCOMES:
Body weight | 12 weeks
Body mass index | 12 weeks
Appendicular skeletal muscle mass index | 12 weeks
  ASMI was measured with a bioimpedance analyser, InBody 270 (InBody, Seoul, South Korea).
6-metre walk test | 12 weeks
  In 6-metre walk test, a 10-metre walkway is marked at the 0-, 2-, 8-, and 10-metre points. The time for the patient to finish the central 6 metres will be recorded by a digital stopwatch by the same tester.
5-time chair stand test | 12 weeks
  Starting from sitting on a standard chair with folded arm across chest, subject is asked to rise from the chair and return to the seated position as quickly as possible for five repetitions.
Short Physical Performance Battery (SPPB) | 12 weeks
  The SPPB, a reliable and valid tool to evaluate functional capability, consisted of three components: standing balance, walking speed and chair stand .

CONTACTS AND LOCATIONS:
Overall Officials: Hin Cheung Leung, MBChB, Principal Investigator — Kowloon Hospital
Locations (1):
- Kowloon Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Zhu LY, Chan R, Kwok T, Cheng KC, Ha A, Woo J. Effects of exercise and nutrition supplementation in community-dwelling older Chinese people with sarcopenia: a randomized controlled trial. Age Ageing. 2019 Mar 1;48(2):220-228. doi: 10.1093/ageing/afy179. PMID 30462162